CLINICAL TRIAL: NCT03395639
Title: An Open-label, Randomised, Parallel-group, Multicentre, Observational Trial to Evaluate Safety and Efficacy of Edoxaban Tosylate in Children From 38 Weeks Gestational Age to Less Than 18 Years of Age With Cardiac Diseases at Risk of Thromboembolic Events
Brief Title: Edoxaban for Prevention of Blood Vessels Being Blocked by Clots (Thrombotic Events) in Children at Risk Because of Cardiac Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DU176b-C-U313; 2017-000475-90 (EudraCT Number)
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Cardiac Disease
Keywords: Children; Pediatrics; Cardiac disease with potential for thromboembolic complications; Prophylactic treatment; Anticoagulant drugs
MeSH Terms: conditions — Heart Diseases | interventions — edoxaban; Standard of Care; Warfarin; Heparin; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Edoxaban (Experimental): Two out of three participants will be randomized for treatment with edoxaban solution or tablets
  Interventions: Drug: Edoxaban
- Standard of Care (SOC) (Active Comparator): One out of three participants will be randomized for treatment with the institution's SOC regimen
  Interventions: Drug: Standard of Care (SOC)

INTERVENTIONS:
Drug: Edoxaban — Edoxaban 15 mg or 30 mg tablets for participants 12 to <18 years of age, or 60 mg edoxaban suspension (dosed as mg/kg) for participants under 12 years of age (and optionally, 12 or older), for oral administration
  Other Names: Lixiana; Savaysa
  Arms: Edoxaban
Drug: Standard of Care (SOC) — Standard of care could include low molecular weight heparin (LMWH) and/or VKA according to the clinical site's SOC treatment regimen
  Other Names: Warfarin/heparin; Enoxaparin
  Arms: Standard of Care (SOC)

SUMMARY:
A committee will judge the safety and effectiveness of edoxaban and the regular treatment (standard of care).

All children in the study will receive free treatment. They will have a 2 in 3 chance to receive edoxaban, and a 1 in 3 chance to receive the standard of care for preventing blood clots.

The study will find out if edoxaban is safer and more effective than the standard of care.

DETAILED DESCRIPTION:
The primary objective is to compare the safety of edoxaban with the standard of care (SOC) in pediatric subjects with cardiac diseases at risk of thromboembolic complications who need primary or secondary anticoagulant prophylaxis with regard to the combination of major and clinically relevant non-major (CRNM) bleeding per International Society on Thrombosis and Haemostasis [ISTH] definition.

The key secondary objective is to compare the efficacy of edoxaban against SOC with regard to the development of symptomatic thromboembolic events (TE) in the systemic arterial or venous pathways including deep vein thrombosis (DVT), pulmonary embolism (PE), stroke, intracardiac thrombus and myocardial infarction (MI), and asymptomatic intracardiac thrombus identified by cardiac imaging.

ELIGIBILITY:
Inclusion Criteria:

* Is a child with cardiac disease who is at risk for thromboembolic complications and requires at least 3 months antithrombotic anticoagulant prophylaxis

Either one of the following:

1. a child with cardiac disease who has a history of cardiac shunt occlusion/thrombosis, with shunt still in place (secondary prevention).

   OR
2. a child with cardiac disease who requires (including those already taking, and those not yet taking) anticoagulation for primary prevention of TE.

Cardiac conditions known to significantly increase the risk of thrombosis (hence, indications for primary TE prevention) are defined in Antithrombotic Therapy and Prevention of Thrombosis. Some examples of cardiac conditions at risk of thrombosis are Fontan surgery, heart failure, Kawasaki disease, and Blalock-Taussig and Glenn surgery.

* Is a male or female child between 1 and <18 years of age (children between 38 weeks gestational age and 1 year of age will be included in the study, however, only after the safety and efficacy data of 50 subjects between 1 and <18 years of age in the edoxaban arm have been evaluated at the end of the 3-month treatment period)
* Has parent(s)/legal guardian(s) or legally acceptable representative who is informed and provides signed consent for the child, to participate in the study with edoxaban treatment. Pediatric participants with appropriate intellectual maturity will be required to sign an assent form in addition to the signed informed consent from the parent(s)/legal guardian(s) or any legally acceptable representative.
* If a female subject of childbearing potential, tests negative for pregnancy at Screening and consents to avoid becoming pregnant by using a locally approved contraception method throughout the study

Exclusion Criteria:

* Has evidence of symptomatic venous or arterial thrombosis and/or asymptomatic intracardiac thrombosis confirmed by a transthoracic echocardiogram during study screening period
* Has mechanical heart valve(s)
* Has active bleeding or high risk of bleeding contraindicating treatment with anticoagulant
* Takes antithrombotic therapy (other than low-dose aspirin) that is not protocol-related
* Administration of rifampin is prohibited during the study and subjects on concomitant use of rifampin are excluded
* Has any hepatic disease associated with coagulopathy leading to a clinically relevant bleeding risk
* Has estimated glomerular filtration rate (eGFR) <30% of normal for age and size
* Has stage 2 hypertension defined as blood pressure systolic and/or diastolic confirmed >99th percentile plus 5 mmHg
* Has thrombocytopenia or life expectancy less than three months
* Has had Fontan procedure with a history of or signs/symptoms suggestive of protein-losing enteropathy
* Is pregnant or breastfeeding
* Has a contraindication to the use of heparin and/or vitamin K antagonist (VKA)
* Has any condition that, as judged by the Investigator, would place the participant at increased risk of harm if he/she participated in the study, including contraindicated medications identified in the protocol

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (48):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cardon Childrens Medical Center, Mesa, Arizona
  - Cedars Sinai Medical Center (ECG), Los Angeles, California
  - University of California-San Francisco Department of Pediatrics - Hematology/Oncology, San Francisco, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Ochsner Medical Center, New Orleans, Louisiana
  - Novant Health Heart and Vascular institute, Charlotte, North Carolina
  - East Carolina Heart Institute @ ECU, Greenville, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - OU Health Sciences Center, Oklahoma City, Oklahoma
  - University of Virginia Health System, Charlottesville, Virginia
  - Seattle Children's Research Institute, Seattle, Washington
- Kepler Universitätsklinikum Med Campus IV, Linz, Austria
- Canada (3):
  - McMaster Children's Hospital, Hamilton, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - McGill University Health Centre/Glen Site/Montreal Children's Hospital, Pierrefonds, Quebec
- University Hospital Center Zagreb, Zagreb, Croatia
- Egypt (5):
  - Zagazig University Hospital, Zagazig, Al Sharkeya
  - Alexandria Clinical Research Center, Faculty of Medicine, Alexandria
  - Kasr Elainy School of Medicine, Abo Elreesh Hospital (Japanese Hospital), Ali Basha Ibrahim ST Faculty of Medicine Cairo University, Cairo
  - Ain Shams University Hospital, Cairo
  - Suez Canal University Hospital, Ismailia
- France (3):
  - Hôpital Des Enfants, Bâtiment Modulaire, Toulouse, Haute Garonne
  - Pediatric and Congenital Cardiology and Pulmonology Department; Arnaud De Villeneuve University Hospital, Montpellier, Herault
  - Pediatric Cardiology Department, Hospital Necker Enfants Malades, APHP, Université Paris Descartes, Paris, Paris Cedex 15
- Hungary (2):
  - Gottsegen Gyorgy Orszagos Kardiologiai Intezet, Budapest
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- India (2):
  - Nirmal Hospital Private Limited, Surat, Gujarat
  - Institute of Child Health, Kolkata
- Israel (3):
  - Soroka University Medical Center, Beersheba
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Lebanon (2):
  - Children's Heart Centre at the American University of Beirut Medical Center, Beirut
  - Hotel Dieu de France Hospital, Beirut
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- Turkey (Türkiye) (5):
  - Erciyes University Medical Faculty, Department of Children Hospital, Edirne, Kayseri
  - Hacettepe University Medical Faculty, Ankara
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Ege University Faculty of Medicine Department of Child Health and Diseases, Izmir
  - Izmir-Dr. Behçet Uz. Pediatric Diseases and Surgery Training and Research Hospital- Izmir Dr. Behcet Uz Cocuk Hastaliklari ve Cerrahisi Egitim ve Arastirma Hastanesi, Izmir
- Ukraine (3):
  - Communal Institution Dnipropetrovsk Regional Pediatric Clinical Hospital of Dnipropetrovsk Regional Council, State Institution Dnipropetrovsk Medical Academy of MoH of Ukraine, Dnipro
  - Communal Healthcare Institution Regional Pediatric Clinical Hospital, Kharkiv National Medical University, Kharkiv
  - Vynnitsa Regional Children Clinical Hospital Policlinic Dept, Vinnytsia
- United Kingdom (3):
  - Royal Brompton Hospital, London, Greater London
  - Glenfield Hospital, Leicester, Leicestershire
  - Ward 2B, Royal Hospital for Children, Glasgow, Strathclyde

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Portman MA, Jacobs JP, Newburger JW, Berger F, Grosso MA, Duggal A, Tao B, Goldenberg NA; ENNOBLE-ATE Trial Investigators. Edoxaban for Thromboembolism Prevention in Pediatric Patients With Cardiac Disease. J Am Coll Cardiol. 2022 Dec 13;80(24):2301-2310. doi: 10.1016/j.jacc.2022.09.031. Epub 2022 Oct 31. PMID 36328157

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 168 participants who met all inclusion criteria and no exclusion criteria were randomized to treatment; 167 participants received treatment and were included in the modified Intent to Treat and Safety Populations.
Pre-assignment Details: All subjects at the Screening Visit were assessed for international normalized ratio (INR) and activated partial thromboplastin time (aPTT) and evaluated at the local laboratory.
Groups:
- Main Treatment Period: Edoxaban; Extension Period: Edoxaban Only: Participants who were randomized to edoxaban solution or tablets orally once a day. Participants 12 to <18 years of age were administered 30 mg, 45 mg, or 60 mg edoxaban tablets or offered granules for oral suspension if they did not have the capacity to swallow. Participants under 12 years of age were administered edoxaban granules (dosed as mg/kg), with maximum dose of 45 mg for 6 months to <12 years, maximum dose of 12 mg for >28 days to <6 months, and maximum dose of 6 mg for 38 weeks gestation to ≤28 days.
- Main Treatment Period: Standard of Care (SOC): Participants who were randomized to SOC regimen which may have included low molecular weight heparin (LMWH) and/or Vitamin K antagonist (VKA) according to the clinical site's SOC treatment regimen.
Period: Main Treatment Period (0 to 4 Months)
Arm/Group | Main Treatment Period: Edoxaban | Main Treatment Period: Standard of Care (SOC) | Extension Period: Edoxaban Only
Started | 110 | 58 | 0
Modified Intent to Treat Population | 109 | 58 | 0
Completed | 107 | 55 | 0
Not Completed | 3 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Participant discontinued at Principal Investigator discretion | 0 | 1 | 0
Period: Extension Period (4-13 Months)
Arm/Group | Main Treatment Period: Edoxaban | Main Treatment Period: Standard of Care (SOC) | Extension Period: Edoxaban Only
Started | 0 | 0 | 147 (15 participants who completed the Main Treatment Period did not participate in the Extension Period)
Completed | 0 | 0 | 144
Not Completed | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Subject discontinued at PI discretion | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Intent to Treat Population (ITT).
Groups:
- Edoxaban: Participants who were randomized to edoxaban solution or tablets orally once a day. Participants 12 to <18 years of age were administered 30 mg, 45 mg, or 60 mg edoxaban tablets or offered granules for oral suspension if they did not have the capacity to swallow. Participants under 12 years of age were administered edoxaban granules (dosed as mg/kg), with maximum dose of 45 mg for 6 months to <12 years, maximum dose of 12 mg for >28 days to <6 months, and maximum dose of 6 mg for 38 weeks gestation to ≤28 days.
- Standard of Care (SOC): Participants who were randomized to SOC regimen which may have included low molecular weight heparin (LMWH) and/or Vitamin K antagonist (VKA) according to the clinical site's SOC treatment regimen.
- Total: Total of all reporting groups
Arm/Group | Edoxaban | Standard of Care (SOC) | Total
Number analyzed (Participants) | 110 | 58 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (4.8) | 7.3 (5.1) | 7.6 (4.9)
Age, Customized [Count of Participants; unit: Participants]
  0 to 6 months | 1 | 3 | 4
  6 months to <2 years | 7 | 5 | 12
  2 to <6 years | 33 | 17 | 50
  6 to <12 years | 41 | 17 | 58
  12 to <18 years | 28 | 16 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 21 | 59
  Male | 72 | 37 | 109
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 3 | 9
  Black or African American | 4 | 3 | 7
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian/Pacific Islander | 2 | 1 | 3
  White | 80 | 39 | 119
  Other | 10 | 7 | 17
  Unknown | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adjudicated Bleeding Events Within the Main Treatment Period
Description: Adjudicated bleeding events included major and clinically-relevant non-major (CRNM) bleeding events per International Society on Thrombosis and Haemostasis (ISTH) definition occurring within the main treatment period. Based on modified ISTH recommendations, major bleeding is defined as a composite (ie, any) of the following: fatal bleeding; and/or symptomatic bleeding in a critical area or organ; and/or bleeding causing a decrease in hemoglobin level of >2 g/dL, or leading to transfusion of the equivalent of ≥2 units of whole blood or red cells. A CRNM bleed is an acute or sub-acute clinically overt bleed that does not meet the criteria for a major bleed but prompts a clinical response, in that it leads to at least one of the following: a hospital admission for bleeding, or a physician guided medical or surgical treatment for bleeding, or a change in antithrombotic therapy. Minor bleeding is any other overt bleeding event that does not meet criteria for either major or CRNM bleeding.
Time Frame: Date of first dose of study drug up to the Month 4 or to the date of last dose of study drug if study treatment was discontinued, whichever was earlier
Population: Adjudicated bleeding events were assessed in participants in the Safety Analysis Set within the Main Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care (SOC)
Number analyzed (Participants) | 109 | 58
Participants
  Major or CRNM bleeding events | 1 | 1
  Major bleeding events | 0 | 0
  All bleeding events (Major, CRNM, minor) | 4 | 2
Statistical Analysis 1: Comparison: Edoxaban vs Standard of Care (SOC); Test type: Other — Difference in adjudicated major or CRNM bleeding rates were assessed; Annualized rate difference = -0.03, 95% CI 2-sided [-0.18 to 0.12]
Statistical Analysis 2: Comparison: Edoxaban vs Standard of Care (SOC); Test type: Other — Difference in adjudicated major bleeding rates were assessed; Annualized rate difference = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 3: Comparison: Edoxaban vs Standard of Care (SOC); Test type: Other — Difference in all adjudicated bleeding (major, CRNM, minor) rates were assessed; Annualized rate difference = 0, 95% CI 2-sided [-0.24 to 0.25]

2. Secondary Outcome: Number of Participants With Symptomatic Thromboembolic Events (TE) in the Systemic Arterial or Venous Pathways Within the Main Treatment Period
Description: Symptomatic thromboembolic events (TE) in the systemic arterial or venous pathways include deep vein thrombosis (DVT), pulmonary embolism (PE), stroke, intracardiac thrombus, and myocardial infarction (MI).
Time Frame: as for outcome 1
Population: Symptomatic thromboembolic events were assessed in participants in the Safety Analysis Set within the Main Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care (SOC)
Number analyzed (Participants) | 109 | 58
Participants
  Thromboembolic event, Any Event | 0 | 1
  Deep vein thrombosis | 0 | 1
  Pulmonary embolism | 0 | 1
  Stroke | 0 | 0
  Systemic embolic event | 0 | 0
  Intracardiac thrombus | 0 | 0
  Myocardial infarction | 0 | 0
  Asymptomatic intracardiac thrombus identified by cardiac imaging | 0 | 0
  Death as a result of TE | 0 | 0

3. Secondary Outcome: Number of Participants Who Died as a Result of Thromboembolic Event Within the Main Treatment Period
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Death was assessed in participants in the modified Intent to Treat Population within the Main Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care (SOC)
Number analyzed (Participants) | 109 | 58
Participants | 0 | 0

4. Secondary Outcome: Number of Participants Who Died as a Result of Any Cause (All-Cause Mortality) Within the Main Treatment Period
Description: Death due to any cause (all-cause mortality) was assessed.
Time Frame: as for outcome 1
Population: Death was assessed in participants in the modified Intent to Treat Population within the Main Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care (SOC)
Number analyzed (Participants) | 109 | 58
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Adjudicated Bleeding Events During the Extension Period
Description: as for outcome 1
Time Frame: Month 4 up to Month 13
Population: Adjudicated bleeding events were assessed in participants with available data in the Safety Analysis Set within the Extension Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban
Number analyzed (Participants) | 144
Participants
  Major or CRNM bleeding events | 1
  Major bleeding events | 1
  All bleeding events (Major, CRNM, minor) | 4

6. Secondary Outcome: Number of Participants With Symptomatic Thromboembolic Events (TE) in the Systemic Arterial or Venous Pathways During the Extension Period
Description: as for outcome 2
Time Frame: Month 4 up to Month 13
Population: Symptomatic thromboembolic events were assessed in participants with available data in the Safety Analysis Set within the Extension Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban
Number analyzed (Participants) | 144
Participants
  Thromboembolic event, Any Event | 4
  Deep vein thrombosis | 0
  Pulmonary embolism | 0
  Stroke | 2
  Systemic embolic event | 0
  Intracardiac thrombus | 0
  Myocardial infarction | 2
  Asymptomatic intracardiac thrombus identified by cardiac imaging | 0
  Death as a result of TE | 0

7. Secondary Outcome: Number of Participants Who Died as a Result of Thromboembolic Event During the Extension Period
Description: as for outcome 2
Time Frame: Month 4 up to Month 13
Population: Death was assessed in participants with available data in the modified Intent to Treat Population within the Extension Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban
Number analyzed (Participants) | 144
Participants | 0

8. Secondary Outcome: Number of Participants Who Died as a Result of Any Cause (All-Cause Mortality) During the Extension Period
Description: Death due to any cause (all-cause mortality) was assessed.
Time Frame: Month 4 up to Month 13
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban
Number analyzed (Participants) | 144
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of signing the informed consent form up to 30 days after the last dose of study drug, up to 13 months.
Description: Adverse events (AEs) were defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Arm/Group | Main Treatment Period: Edoxaban | Main Treatment Period: Standard of Care (SOC) | Extension Period: Edoxaban Only
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/58 | 2/144
Serious Adverse Events (participants affected / at risk) | 5/109 | 3/58 | 19/144
Other Adverse Events (participants affected / at risk) | 51/109 | 24/58 | 69/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Treatment Period: Edoxaban (N=109) | Main Treatment Period: Standard of Care (SOC) (N=58) | Extension Period: Edoxaban Only (N=144)
Cardiac failure (Cardiac disorders) | 2 | 1 | 0
Coronary artery thrombosis (Cardiac disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Coarctation of the aorta (Congenital, familial and genetic disorders) | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 2
Abscess limb (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pulmonary arterial pressure increased (Investigations) | 0 | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Treatment Period: Edoxaban (N=109) | Main Treatment Period: Standard of Care (SOC) (N=58) | Extension Period: Edoxaban Only (N=144)
Bronchitis (Infections and infestations) | 3 | 0 | 3
Pyrexia (General disorders) | 5 | 1 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 2 | 9
Headache (Nervous system disorders) | 5 | 2 | 9
Iron deficiency (Metabolism and nutrition disorders) | 0 | 2 | 0
Catheterisation cardiac (Investigations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 7
Nasopharyngitis (Infections and infestations) | 4 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3
Influenza (Infections and infestations) | 1 | 0 | 5
Tonsillitis (Infections and infestations) | 2 | 0 | 3
Viral infection (Infections and infestations) | 0 | 1 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Haematoma (Vascular disorders) | 0 | 0 | 5
Laryngitis (Infections and infestations) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT03395639/Prot_SAP_000.pdf